CLINICAL TRIAL: NCT00035763
Title: Pain in Sickle Cell Epidemiologic Study
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1105; R01HL064122 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2008-01

CONDITIONS: Blood Disease; Anemia, Sickle Cell
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell

SUMMARY:
To measure the variability in pain and response to pain in sickle cell disease, and to build multivariate models to explain both patients' pain and their response to pain, especially, utilization of health care.

DETAILED DESCRIPTION:
BACKGROUND:

Pain in sickle cell disease is poorly recognized, measured, and treated. Although painful episodes are the most common reason sickle cell patients seek care, studies have seldom directly measured pain in detail. In studies to date, biological and demographic variables alone only partly explain the observed variance in painful episode frequency. Further, little is known about differences in pain responses including home management versus health care utilization.

DESIGN NARRATIVE:

This cohort study is measuring the variability in pain and response to pain in sickle cell disease, and building multivariate models to explain both patients' pain and their response to pain, especially, utilization of health care. The models' outcome variables include mean pain, painful episodes, and various types of utilization episodes, including non-narcotic analgesic use, narcotic use, office visits, emergency department (ED visits, and hospitalization. An additional outcome is the percentage of each patient's painful episodes that result in various types of utilization. Outcomes will be operationalized using daily pain diaries collected over six months. Reflecting on the prior 24 hours, patients will recall on an ordinal (0-9) scale maximum pain, distress, and disability, judge whether they were in a "crisis," and note pain locations and their various types of utilization. Daily pain intensity ratings will be transformed into pain episode counts using a formulaic threshold for a painful episode. The formula calculates each patient's threshold individually, based on his/her pain ratings. The models will measure the effect of several classes of explanatory variables (demographic, disease-related, psycho social, and readiness to utilize care), operationalized using primary data and validated instruments.

Patients will be recruited from the central and Tidewater regions of Virginia, will undergo an initial survey battery, chart review, and a brief final survey, venipuncture and urine sampling, and complete pain diaries daily for six months. This study will advance knowledge of the etiology and influences on pain and pain response in sickle cell disease. By revealing potentially mutable explanatory variables, the study's results will suggest targets of biobehavioral treatment interventions.

ELIGIBILITY:
No eligibility criteria

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wally Smith — Virginia Commonwealth University

REFERENCES:
- [Background] Smith WR, Bovbjerg VE, Penberthy LT, McClish DK, Levenson JL, Roberts JD, Gil K, Roseff SD, Aisiku IP. Understanding pain and improving management of sickle cell disease: the PiSCES study. J Natl Med Assoc. 2005 Feb;97(2):183-93. PMID 15712781